CLINICAL TRIAL: NCT04538976
Title: Copd Exacerbation and Pulmonary Hypertension Trial
Acronym: CODEX-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study_protocol_CODEX-P_ver2_1
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Acute Exacerbation of COPD
Keywords: COPD; Chronic Obstructive Lung Disease; Increased pulmonary pressure; Acute Exacerbation; AECOPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: The study is a multicenter controlled, randomized, open-lapel trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients in the control group will receive standard care.
- Sildenafil (Active Comparator): Patients in the Sildenafil group will receive standard care and targeted Sildenafil-treatment.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil in standard dosage
  Other Names: Vizarsin
  Arms: Sildenafil

SUMMARY:
This trial will investigate whether patiens admitted with an acute exacerbation of chronic obstructive lung disease and pulmonary hypertension will benefit from a targeted pharmacological treatment.

DETAILED DESCRIPTION:
During admittance due to acute exacerbation of chronic obstructive lung disease will patience have an echocardiography to examine their pulmonary pressure. If patient have a tricuspidal return gradient above 40 mmHg, they will receive treatment with a phosphordiesterase-5-inhibitor, Sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* COPD verified by specialist and spirometry
* Admitted with the diagnosis "acute exacerbation of COPD"
* TR-gradient ≥40 mmHg verified by specialist and echocardiography
* Informed consent

Exclusion Criteria:

* Known pulmonal hypertension
* Known heart disease which affects the pump function of the heart
* Men <40 years
* Women <55 years
* Not-menopauseal women <55 years (Menopause is defined as no menstruation within 12 months.)
* Severe mental illness which significantly complicates cooperation
* Severe language difficulties which significantly complicates cooperation
* known allergy to Sildenafil
* Sildenafil consumption ≥50 mg / week due to other indications

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Time alive and out of hospital | 365 days

SECONDARY OUTCOMES:
Time to "prednisolon and/or antibiotica"-needing exacerbation of COPD or death | 365 days
Death within 90 days | 90 days
Death within 1 year | 365 days
Alive and without exacerbation of COPD on day 365 | 365 days
Clinical cure | 14 days
Number of readmissions due to exacerbations of COPD | 365 days
Number of days with non-invasive ventilation (NIV) or respirator during admittance | 14 days
Delta Pa(O2) | 4 days
Delta Pa(CO2) | 4 days
Delta(pH) | 4 days
Change in FEV1 | 90 days
Change in COPD Assesment Test (CAT) | 29 days
Change in Body Mass Index (BMI) | 90 days
Delta(TR-gradient) | 4 days

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Bispebjerg University Hospital, Copenhagen
  - Herlev-Gentofte Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Nordsjællands Hospital, Hillerød
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: No
We have not yet decided to share IPD.